CLINICAL TRIAL: NCT04771741
Title: Opiate Free Multimodal Pain Pathway in Elective Foot and Ankle Surgery: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Prisma Health-Midlands (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00099067
Record Dates: First submitted 2021-02-18; First posted 2021-02-25 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Bunion of Unspecified Foot; Bunionette of Unspecified Foot; Hammertoe; Ankle Fractures; Achilles Tendon Surgery
MeSH Terms: conditions — Hammer Toe Syndrome; Ankle Fractures | interventions — Acetaminophen; Ketorolac Tromethamine; Ketorolac; Meloxicam; cyclobenzaprine; Pregabalin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Multimodal Pain Pathway: This group will receive the multimodal pain pathway cocktail of medications. This cocktail includes:
  * Tylenol (acetominophen), 1000 mg, every 6 hours as needed for pain
  * Ketorolac (Toradol), 10 mg, every 6 hours as needed for pain until post-op day 3
  * Mobic (Meloxicam), 15 mg once daily, beginning on post-op day 4
  * Flexeril (Cyclobenzaprine), 10 mg every 8 hours as needed for pain
  * Pregabalin (Lyrica), 75 mg every 12 hours as needed for pain
  Interventions: Drug: Acetominophen; Drug: Toradol; Drug: Meloxicam; Drug: Cyclobenzaprine; Drug: Lyrica

INTERVENTIONS:
Drug: Acetominophen — 1,000 mg every 6 hours
  Other Names: Tylenol
Drug: Toradol — 10 mg every 6 hours, days 0-3
  Other Names: Ketorolac
Drug: Meloxicam — 15 mg once daily, beginning post-op day 4
  Other Names: Mobic
Drug: Cyclobenzaprine — 10 mg every 8 hours
  Other Names: Flexeril
Drug: Lyrica — 75 mg every 12 hours
  Other Names: Pregabalin

SUMMARY:
Orthopedic surgeons frequently prescribe and over-prescribe narcotic pain medications during the postoperative period, despite the ongoing opioid crisis in the United States. While opioid-free multimodal pathways have shown promising results, there remains a lack of published literature evaluating opiate-free multimodal pain protocols for elective outpatient foot and ankle surgeries. This study aims to evaluate post-operative pain following the use of an opioid-free pain treatment plan for patients undergoing foot and ankle surgeries.

DETAILED DESCRIPTION:
Despite the presence and increased understanding of the opioid crisis in the United States, orthopedic surgeons frequently prescribe and over-prescribe narcotic pain medications during the postoperative period. In an effort to minimize narcotic analgesia and its potential side effects, opioid-free multimodal pathways have been developed in many orthopaedic sub-specialties with promising results. There have been early studies reporting the results of non-narcotic protocols during the intra-operative period. Likewise, there have been several studies reporting the results of inpatient non-narcotic pain protocols in select foot and ankle surgeries. However, there remains a lack of published literature evaluating opiate-free multimodal pain protocols for elective outpatient foot and ankle surgeries. Currently, our practice utilizes an opioid-free post-operative pain protocol for patients undergoing elective outpatient foot and ankle surgery. The goal of this study is to evaluate post-operative pain using this opioid-free multimodal pain protocol at days 1,3, and 8 following elective outpatient foot and ankle surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Outpatient, elective, primary foot and ankle surgery not due to infection including:
* Bunion or bunionette surgery, hammertoe surgery, ankle fracture, Achilles tendon surgery (primary mid-substance repair, Haglund's deformity correction with debridement), ankle arthroscopy

Exclusion Criteria:

* <18 years of age
* Undergoing revision surgery
* Allergic to more than 1 medication listed in protocol
* Creatinine clearance >1.5
* Known end-stage renal, stage 2 or higher
* History of GI bleed, ulcer, NSAID-induced gastritis, and/or gastric bypass
* History of active liver disease or Child-Pugh Class 2 liver failure or above
* History of pain syndromes including: fibromyalgia, complex regional pain syndrome/reflex sympathetic dystrophy, hyperalgesia
* Inability to undergo regional anesthesia due to inability to obtain nerve block, prior nerve damage or anatomy, or anesthesiologic best judgement
* Currently pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included in this study will be adult outpatient, elective, primary foot and ankle surgery that is not due to infection performed at Prisma Health Orthopedics.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with opioid-free multimodal postoperative protocol. | 2 weeks
  Study participants will complete a survey at the 2 week follow-up visit asking yes or no if they were satisfied with the opioid-free pain management protocol.
Rate of failure of opioid-free multimodal postoperative protocol. | 2 weeks
  At 2 weeks, patients will be asked yes or no if they used any additional medications for pain outside of prescriptions that were provided in the opioid-free multimodal pain protocol.

SECONDARY OUTCOMES:
Post-operative Pain: Day 1 | 1 day
  Study participants will be asked to rate their pain using a Visual Analog Scale (VAS) from 0 (no pain) to 10 (worst pain) at post-operative day 1.
Post-operative Pain: Day 3 | 3 days
  Study participants will be asked to rate their pain using a Visual Analog Scale (VAS) from 0 (no pain) to 10 (worst pain) at post-operative day 3.
Post-operative Pain: Day 8 | 8 days
  Study participants will be asked to rate their pain using a Visual Analog Scale (VAS) from 0 (no pain) to 10 (worst pain) at post-operative day 8.

CONTACTS AND LOCATIONS:
Overall Officials: J. Benjamin Jackson, MD, MBA, Principal Investigator — Prisma Health-Midlands
Locations (1):
- Prisma Health Midlands, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haddad DK, Sherman OH. Developing opioid prescribing recommendations in the postoperative orthopedic setting. J Opioid Manag. 2019 Jul/Aug;15(4):333-341. doi: 10.5055/jom.2019.0518. PMID 31637685
- [Background] Janakiram C, Fontelo P, Huser V, Chalmers NI, Lopez Mitnik G, Brow AR, Iafolla TJ, Dye BA. Opioid Prescriptions for Acute and Chronic Pain Management Among Medicaid Beneficiaries. Am J Prev Med. 2019 Sep;57(3):365-373. doi: 10.1016/j.amepre.2019.04.022. Epub 2019 Aug 1. PMID 31377093
- [Background] Young JD, Bhashyam AR, Qudsi RA, Parisien RL, Shrestha S, van der Vliet QMJ, Fils J, Losina E, Dyer GSM. Cross-Cultural Comparison of Postoperative Discharge Opioid Prescribing After Orthopaedic Trauma Surgery. J Bone Joint Surg Am. 2019 Jul 17;101(14):1286-1293. doi: 10.2106/JBJS.18.01022. PMID 31318808
- [Background] Bean BA, Connor PM, Schiffern SC, Hamid N. Outpatient Shoulder Arthroplasty at an Ambulatory Surgery Center Using a Multimodal Pain Management Approach. J Am Acad Orthop Surg Glob Res Rev. 2018 Oct 23;2(10):e064. doi: 10.5435/JAAOSGlobal-D-18-00064. eCollection 2018 Oct. PMID 30656252
- [Background] Seki H, Ideno S, Ishihara T, Watanabe K, Matsumoto M, Morisaki H. Postoperative pain management in patients undergoing posterior spinal fusion for adolescent idiopathic scoliosis: a narrative review. Scoliosis Spinal Disord. 2018 Sep 12;13:17. doi: 10.1186/s13013-018-0165-z. eCollection 2018. PMID 30214945
- [Background] Garcia RM, Cassinelli EH, Messerschmitt PJ, Furey CG, Bohlman HH. A multimodal approach for postoperative pain management after lumbar decompression surgery: a prospective, randomized study. J Spinal Disord Tech. 2013 Aug;26(6):291-7. doi: 10.1097/BSD.0b013e318246b0a6. PMID 23887076
- [Background] Seiter M, Aiyer A. Current Trends in Anesthesia Management in Hallux Valgus. Foot Ankle Clin. 2020 Mar;25(1):47-57. doi: 10.1016/j.fcl.2019.10.002. Epub 2019 Nov 20. PMID 31997746
- [Background] Lee JK, Kang C, Hwang DS, Lee GS, Hwang JM, Park EJ, Ga IH. An Innovative Pain Control Method Using Peripheral Nerve Block and Patient-Controlled Analgesia With Ketorolac After Bone Surgery in the Ankle Area: A Prospective Study. J Foot Ankle Surg. 2020 Jul-Aug;59(4):698-703. doi: 10.1053/j.jfas.2019.12.001. Epub 2020 Feb 10. PMID 32057624
- [Background] Michelson JD, Addante RA, Charlson MD. Multimodal analgesia therapy reduces length of hospitalization in patients undergoing fusions of the ankle and hindfoot. Foot Ankle Int. 2013 Nov;34(11):1526-34. doi: 10.1177/1071100713496224. Epub 2013 Jul 8. PMID 23836812
- [Background] McDonald EL, Daniel JN, Rogero RG, Shakked RJ, Nicholson K, Pedowitz DI, Raikin SM, Bilolikar V, Winters BS. How Does Perioperative Ketorolac Affect Opioid Consumption and Pain Management After Ankle Fracture Surgery? Clin Orthop Relat Res. 2020 Jan;478(1):144-151. doi: 10.1097/CORR.0000000000000978. PMID 31567579